CLINICAL TRIAL: NCT00058838
Title: A Phase III, Double-Blind, Placebo-Controlled, Fixed-Dose Response Study Comparing the Efficacy and Safety of Sumanirole Versus Placebo in Patients With Early Parkinson's Disease.
Brief Title: Study Evaluating Sumanirole for the Treatment of the Signs and Symptoms of Early Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DA2APD-0075-031
Record Dates: First submitted 2003-04-14; First posted 2003-04-15 (Estimated); Last update posted 2006-06-07 (Estimated); Status verified 2006-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — U 95666E

INTERVENTIONS:
Drug: sumanirole

SUMMARY:
The primary purpose of this study is to determine whether sumanirole, at three different dose levels, is effective and safe in the treatment of the signs and symptoms of early Parkinson's disease

ELIGIBILITY:
Inclusion Criteria:

Idiopathic Parkinson's disease < 7 years duration

Modified Hoehn and Yahr Scale Stages I through III

Age greater than or equal to 30 years old

Patients or their partners must use adequate contraceptive methods

Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures and do not plan on traveling extensively during the study

Exclusion Criteria:

Atypical Parkinson's disease syndromes due to drugs, metabolic disorders, encephalitis, or degenerative diseases.

Levodopa received for 1-year accumulated interval in the last two years.

Dopamine agonist medications or catechol-o-methyl transferase inhibitors in the 30 days prior to baseline.

Unstable dose regimes of hypnotics, anxiolytics or antidepressants

Dementia

History of stereotaxic brain surgery, psychosis or active epilepsy within past year.

Participation in clinical trial within the previous 30 days.

Malignant melanoma or history of melanoma

Significant medical or pshychiatric condition

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 854
Dates: Start 2003-04; Study Completion 2004-09

PRIMARY OUTCOMES:
Change from baseline in UPDRS (Unified Parkinson's Disease Rating Scale) II + III total scores at end of maintenance, for sumanirole compared to placebo

SECONDARY OUTCOMES:
To assess the safety profile of sumanirole and the benefit of sumanirole in quality of life measures compared to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (117):
- United States (63):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Concord, California
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Loma Linda, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, Oxnard, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, Sunnyvale, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Englewood, Colorado
  - Pfizer Investigational Site, Fort Collins, Colorado
  - Pfizer Investigational Site, Fairfield, Connecticut
  - Pfizer Investigational Site, Hartford, Connecticut
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Maitland, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Palm Beach Gardens, Florida
  - Pfizer Investigational Site, Sarasota, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Tallahasse, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Marietta, Georgia
  - Pfizer Investigational Site, Savannah, Georgia
  - Pfizer Investigational Site, Elkhart, Indiana
  - Pfizer Investigational Site, Des Moines, Iowa
  - Pfizer Investigational Site, Dubuque, Iowa
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Southfield, Michigan
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Canfield, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Dayton, Ohio
  - Pfizer Investigational Site, Bend, Oregon
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, Upland, Pennsylvania
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Tacoma, Washington
  - Pfizer Investigational Site, Wenatchee, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Argentina (2):
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires F.D.
- Australia (5):
  - Pfizer Investigational Site, Sydney, New South Wales
  - Pfizer Investigational Site, Westmead, New South Wales
  - Pfizer Investigational Site, Herston, Queensland
  - Pfizer Investigational Site, Adelaide, South Australia
  - Pfizer Investigational Site, Nedlands, Western Australia
- Austria (4):
  - Pfizer Investigational Site, Innsbruck
  - Pfizer Investigational Site, Linz
  - Pfizer Investigational Site, Sankt Pölten
  - Pfizer Investigational Site, Vienna
- Belgium (5):
  - Pfizer Investigational Site, Antwerp
  - Pfizer Investigational Site, Edegem
  - Pfizer Investigational Site, Ottignies
  - Pfizer Investigational Site, Roeselaere
  - Pfizer Investigational Site, Tielt
- Colombia (2):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Bogotá, D.C.
- France (5):
  - Pfizer Investigational Site, Aix-en-Provence
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Montbelliard
  - Pfizer Investigational Site, Nîmes
  - Pfizer Investigational Site, Roanne
- Germany (4):
  - Pfizer Investigational Site, Gera
  - Pfizer Investigational Site, Hamburg
  - Pfizer Investigational Site, Straubing
  - Pfizer Investigational Site, Wiesbaden
- Greece (2):
  - Pfizer Investigational Site, Athens, Attica
  - Pfizer Investigational Site, Thessaloniki, Macedonia
- Italy (8):
  - Pfizer Investigational Site, Lido di Camaiore, LU
  - Pfizer Investigational Site, Florence
  - Pfizer Investigational Site, Grosseto
  - Pfizer Investigational Site, Imperia
  - Pfizer Investigational Site, Milan
  - Pfizer Investigational Site, Napoli
  - Pfizer Investigational Site, Pozzilli
  - Pfizer Investigational Site, Torino
- Mexico (3):
  - Pfizer Investigational Site, Mexico City, D.F.
  - Pfizer Investigational Site, Zapopan, Jalisco
  - Pfizer Investigational Site, Mexico City, Mexico City
- Pfizer Investigational Site, Lima, Lima Province, Peru
- Puerto Rico (2):
  - Pfizer Investigational Site, Carolina
  - Pfizer Investigational Site, Ponce
- Spain (11):
  - Pfizer Investigational Site, Ávila, Avila
  - Pfizer Investigational Site, Barcelona, Barcelona
  - Pfizer Investigational Site, Terrassa, Barcelona
  - Pfizer Investigational Site, Donostia / San Sebastian, Guipuzcoa
  - Pfizer Investigational Site, Alcalá de Henares, Madrid
  - Pfizer Investigational Site, Madrid, Madrid
  - Pfizer Investigational Site, Oviedo, Oviedo
  - Pfizer Investigational Site, Barcelona
  - Pfizer Investigational Site, Burgos
  - Pfizer Investigational Site, Madrid
  - Pfizer Investigational Site, Zaragoza

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=DA2APD-0075-031&StudyName=Study+evaluating+sumanirole+for+the+treatment+of+the+signs+and+symptoms+of+early+Parkinson%27s+disease